CLINICAL TRIAL: NCT01838473
Title: In-vivo Extraction of Lead, Cadmium and Tobacco Specific Nitrosamines From Four Brands of Swedish 'Snus' in Regular Snus Users.
Brief Title: In-vivo Extraction of Lead, Cadmium and Tobacco Specific Nitrosamines From Swedish 'Snus' in Regular Snus Users
Acronym: SMWS03
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Contract Research Organization el AB (Industry)
Collaborators: Swedish Match AB (Industry)
Responsible Party: Principal Investigator, Erik Lunell, MD, PhD, MD, PhD, Contract Research Organization el AB
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: SMWS03
Record Dates: First submitted 2012-02-10; First posted 2013-04-24 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Smoking Cessation; Harm Reduction
Keywords: smokeless tobacco; Nicotine; Cadmium; lead; Tobacco Specific Nitrosamines
MeSH Terms: conditions — Smoking Cessation; Harm Reduction; Tobacco Use | interventions — Tobacco, Smokeless

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- General 1 g pouch (Active Comparator): Oral pouch 0.3-1g, single dose. One pouch administered over 30 minutes. Buccal Administration of nicotine.
  Interventions: Procedure: Buccal Administration of nicotine
- Catch Licoice 1 g pouch (Active Comparator): Oral pouch 1g, single dose. One pouch administered over 30 minutes. Buccal Administration of nicotine.
  Interventions: Procedure: Buccal Administration of nicotine
- Catch Licorice Mini 0.5 g pouch (Active Comparator): Oral pouch 0.5g, single dose. One pouch administered over 30 minutes. Buccal Administration of nicotine.
  Interventions: Procedure: Buccal Administration of nicotine
- Catch Licorice dry mini 0.3 g pouch (Active Comparator): Oral pouch 0.3 g, single dose. One pouch administered over 30 minutes. Buccal Administration of nicotine.
  Interventions: Procedure: Buccal Administration of nicotine

INTERVENTIONS:
Procedure: Buccal Administration of nicotine — Oral pouch 1g, single dose. One pouch administered over 30 minutes.
  Other Names: Smokeless tobacco; ST; Potential Exposure Reduced Product; PREP
  Arms: General 1 g pouch
Procedure: Buccal Administration of nicotine — Oral pouch 1g, single dose. One pouch administered over 30 minutes.
  Other Names: Smokeless tobacco; ST; Potential Exposure Reduced Product; PREP
  Arms: Catch Licoice 1 g pouch
Procedure: Buccal Administration of nicotine — Oral pouch 0.5 g, single dose. One pouch administered over 30 minutes.
  Other Names: Smokeless tobacco; ST; Potential Exposure Reduced Product; PREP
  Arms: Catch Licorice Mini 0.5 g pouch
Procedure: Buccal Administration of nicotine — Oral pouch 0.3 g, single dose. One pouch administered over 30 minutes.
  Other Names: Smokeless tobacco; ST; Potential Exposure Reduced Product; PREP
  Arms: Catch Licorice dry mini 0.3 g pouch

SUMMARY:
In an open label, randomized, two-way cross-over study, 32 male healthy regular snus users will be given repeated doses of four different types of portion snus: "General", "Catch", "Catch Mini" and "Catch Dry Mini". Each portion of used snus will be collected and frozen (-20 oC) pending analysis of lead (Pb), cadmium (Cd), nicotine and tobacco specific nitrosamines (TSNAs). Unused snus is collected and deep frozen for analysis and calculation of extracted dose. Calculations of extracted amount of lead, cadmium, nicotine and tobacco specific nitrosamines (TSNAs) respectively, will be done for each type of snus.

DETAILED DESCRIPTION:
Comparisons:

A= "General Portion" 1 g portion snus containing approximately 8 mg nicotine per portion.

B= "Catch Licorice Portion" 1 g portion snus containing approximately 8 mg nicotine per portion.

C= "Catch Licorice Portion Mini" 0.5 g portion snus containing approximately 4 mg nicotine per portion.

D= "Catch Dry Licorice Portion Mini" 0.3 g portion snus containing approximately 4 mg nicotine per portion.

Swedish portion snus will be administered once every hour (4 administrations/brand) and will be kept between the upper lip and the gum for 30 minutes. Preload of own brand each morning.

ELIGIBILITY:
Inclusion Criteria:

* non-smokers, 18 to 50 years of age.
* Habitual use of > 7 portions snus daily since minimum 1 year.
* Healthy according to the health declaration and interview.
* Written informed consent given.

Exclusion Criteria:

* Concurrent participation in another clinical trial.
* History of allergy.
* History of allergy.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2004-05; Primary Completion 2004-08 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
In-vivo extraction of cadmium | 30 minutes' use
  Extracted amount = mean of 10 unused sachets - residual amount

SECONDARY OUTCOMES:
in-vivo extraction of tobacco specific nitrosamines (TSNAs) | 30 minutes' use
  Extracted amount = mean of 10 unused sachets - residual amount in used sachet
In-vivo extraction of lead | 30 minutes' use
  Extracted amount = mean of 10 unused sachets - residual amount in one used sachet
In-vivo extraction of nicotine | 30 minutes' use
  Extracted amount = mean of 10 unused sachets - residual amount in one used sachet

CONTACTS AND LOCATIONS:
Overall Officials: Erik Lunell, MD, PhD, Principal Investigator — Croel AB
Locations (1):
- CROel AB, Helsingborg, Sweden